CLINICAL TRIAL: NCT06735118
Title: Feasibility Study of Deep Learning-based MDixon Quant for Quantitative Assessment of Chemotherapy-induced Fatty Liver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: KYLX2023-165
Record Dates: First submitted 2024-11-27; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- neoadjuvant chemotherapy group (Experimental): Cancer patients undergoing chemotherapy.
  Interventions: Drug: Neoadjuvant chemotherapy
- Non-neoadjuvant chemotherapy group (No Intervention): Cancer patients not undergoing chemotherapy.

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Neoadjuvant chemotherapy
  Other Names: Non
  Arms: neoadjuvant chemotherapy group

SUMMARY:
The purpose of this study is to quantitatively assess the changes in liver fat content in cancer patients before and after treatment.

The main questions it aims to answer are:How does the liver fat fraction change before and after chemotherapy? In this study, patients undergoing mDixon Quant scanning are subjected to fully automated segmentation and measurement of liver fat content using artificial intelligence.

DETAILED DESCRIPTION:
Regarding the extraction of liver fat fraction, the traditional axial ROI method involves selecting several regions of interest (ROIs) at the largest cross-sectional level or across multiple continuous sections, and taking the average value as the whole-liver fat fraction. This method is complex, time-consuming, and cannot obtain the whole-liver fat fraction. In this study, a threshold extraction method is used to obtain the whole-liver fat fraction, enabling a 2D-to-3D conversion, which is more time-efficient and labor-saving, and provides a more accurate measurement.

ELIGIBILITY:
Inclusion Criteria:

1. CT/B ultrasound showed no fatty liver
2. No MRI contraindications, including pacemaker, stent, metal implant, or claustrophobia
3. Received neoadjuvant/adjuvant chemotherapy

Exclusion Criteria:

1. Missing follow-up information
2. Liver lesions (metastases, hemangioma, etc.)
3. Poor image quality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Extract the whole liver fat fraction | one year
  Extract the whole liver fat fraction using the threshold extraction method.

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — Ethics Committee of Yunnan Provincial Cancer Hospital
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No